CLINICAL TRIAL: NCT06953037
Title: Effects of Acupressure Applied Before Cesarean Delivery on Anxiety, Physiological Parameters and Fetal Heart Rate: A Randomized Controlled Trial
Brief Title: Effects of Acupressure Applied Before Cesarean Delivery on Anxiety, Physiological Parameters and Fetal Heart Rate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Arzu Abiç, Asist Prof Dr, Eastern Mediterranean University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: ETK00-2024-0222; EASTERN MEDİTERRANEAN UNI (Other: EASTERN MEDİTERRANEAN UNI)
Record Dates: First submitted 2025-03-12; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Caesarean Section; Pregnant Women; Anxiety Disorder
Keywords: pregnant women; caesarean section; anxiety; fetal heart rate; accupressure
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupressure (Experimental): The acupressure points to be used in the study are the San Yin Jiao points on the spleen meridian (SP6) located on the inside of the lower leg, 4 fingers above the ankle and behind the tibia, which are effective in reducing anxiety, and the Shen Men points on the heart meridian (HT7) located in the small pit between the pisiform and ulna (elbow) bones in the transverse wrist fold. Acupressure will be applied to the women in the acupressure group by a certified researcher.
  Interventions: Other: acupressure
- control (No Intervention): routine nursing care

INTERVENTIONS:
Other: acupressure — The application will be made to the women in the acupressure group after applying the data collection forms (Personal Information Form, STAI-1 and Physiological Parameters and Fetal Heart Rate Chart) 1 hour before the cesarean section. The application will be made to the women in the acupressure group by manually pressing the SP6 and HT7 points with the index or middle finger for 5 seconds to a depth of 1-1.5 cm in the order determined by lot, then resting for 2 seconds and continuing the application for 2 minutes. Anxiety, physiological parameters and fhr will be measured again 40 minutes after the application. The data collection forms (descriptive characteristics form, loss, physiological parameters, fhr) will be applied to the women in the control group 1 hour before the cesarean section. No intervention will be made to the women in the control group. Anxiety, physiological parameters and fhr will be measured again 40 minutes later.
  Arms: acupressure

SUMMARY:
Cesarean section is the most commonly preferred surgical method in cases where vaginal birth is not possible or complications that may endanger the health of the mother and baby occur. Cesarean section rates are increasing worldwide. According to the latest data (2010-2018) from 154 countries covering 94.5% of live births in the world, 21.1% of women have cesarean section births and it is estimated that this rate will increase to 28.5% by 2030. According to the Centers for Disease Control and Prevention (CDC), the cesarean section rate in the USA, which was 32.1% in 2022, increased to 32.4% in 2023. When the cesarean section rates of the Turkey Demographic Health Survey (TDHS) are examined, the rate, which was 7% in 1993, increased to 52% in 2018, an increase of 45% is observed. In the TRNC, this rate was 11.1% in 1981, but in 2017 this rate increased by an average of 7 times, reaching 72.5%. Pregnant women tend to have cesarean sections because they are affected by the risks that will occur during birth, negative birth stories told among the public, and painful birth scenes seen on social media. Studies have shown that despite the high rates of cesarean sections in pregnant women's birth methods, a significant increase in women's anxiety levels is observed. While waiting for the surgery, pre-operative anxiety, fear of the procedure, etc. are more common than other feelings and symptoms.Studies have also shown that anxiety increases in patient rooms, the night before surgery, and when moving to the operating table. In a study conducted by Lopez, the most important causes of preoperative anxiety were listed as fear of the hospital environment (35%), fear of surgery (33%), fear of anesthesia (45%), and unawareness of the surgery (45%). Concerns about the success of the operation (29.3%), fear of postoperative prognosis (19.5%), and surgical complications (11.4%) are the most common causes of preoperative anxiety. High levels of anxiety experienced before surgery cause increased heart rate, blood pressure, and oxygen consumption during surgery.

Controlling and managing preoperative anxiety is one of the most important goals of nursing care worldwide, as in cesarean cases. Mothers need to relax mentally and physically after cesarean sections so that they can care for their babies after birth. A common way to control preoperative anxiety is to use sedatives, but these medications can cause side effects. Therefore, acupressure, which is a non-invasive, low-cost, uncomplicated and non-pharmacological method due to fewer complications, can be used to reduce preoperative anxiety. Acupressure is the application of pressure to stimulate acupoints and meridian lines using an object or fingers, without the use of needles. Acupressure is a simple treatment approach and can be applied by nurses or patients who have received the necessary training, because it is simple and does not require any equipment.

DETAILED DESCRIPTION:
Cesarean section is the most commonly preferred surgical method in cases where vaginal birth is not possible or complications that may endanger the health of the mother and baby occur. Cesarean section rates are increasing worldwide. According to the latest data (2010-2018) from 154 countries covering 94.5% of live births in the world, 21.1% of women have cesarean section births and it is estimated that this rate will increase to 28.5% by 2030. According to the Centers for Disease Control and Prevention (CDC), the cesarean section rate in the USA, which was 32.1% in 2022, increased to 32.4% in 2023. When the cesarean section rates of the Turkey Demographic Health Survey (TDHS) are examined, the rate, which was 7% in 1993, increased to 52% in 2018, an increase of 45% is observed. In the TRNC, this rate was 11.1% in 1981, but in 2017 this rate increased by an average of 7 times, reaching 72.5%. Pregnant women tend to have cesarean sections because they are affected by the risks that will occur during birth, negative birth stories told among the public, and painful birth scenes seen on social media. Studies have shown that despite the high rates of cesarean sections in pregnant women's birth methods, a significant increase in women's anxiety levels is observed. While waiting for the surgery, pre-operative anxiety, fear of the procedure, etc. are more common than other feelings and symptoms.Studies have also shown that anxiety increases in patient rooms, the night before surgery, and when moving to the operating table. In a study conducted by Lopez, the most important causes of preoperative anxiety were listed as fear of the hospital environment (35%), fear of surgery (33%), fear of anesthesia (45%), and unawareness of the surgery (45%). Concerns about the success of the operation (29.3%), fear of postoperative prognosis (19.5%), and surgical complications (11.4%) are the most common causes of preoperative anxiety. High levels of anxiety experienced before surgery cause increased heart rate, blood pressure, and oxygen consumption during surgery.

Controlling and managing preoperative anxiety is one of the most important goals of nursing care worldwide, as in cesarean cases. Mothers need to relax mentally and physically after cesarean sections so that they can care for their babies after birth. A common way to control preoperative anxiety is to use sedatives, but these medications can cause side effects. Therefore, acupressure, which is a non-invasive, low-cost, uncomplicated and non-pharmacological method due to fewer complications, can be used to reduce preoperative anxiety. Acupressure is the application of pressure to stimulate acupoints and meridian lines using an object or fingers, without the use of needles. Acupressure is a simple treatment approach and can be applied by nurses or patients who have received the necessary training, because it is simple and does not require any equipment.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study,
* Be between the ages of 18-45,
* Have a caesarean section between 37-40 weeks,
* Not have a risky pregnancy,
* Have spinal anesthesia,

Exclusion Criteria:

* Not having anxiety 1 hour before the cesarean section,
* Having a risky pregnancy,
* Having a chronic disease,
* Having a severe systemic disease,
* Not receiving spinal anesthesia,
* Having a body mass index over 25,
* Having previous acupressure experience,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Scale | 1 DAY
  The state anxiety scale was developed by Spielberg et al. (1970) and adapted to Turkish by Öner and Le Compte (1983). The State Anxiety Scale, which was developed to measure an individual's anxiety at a certain moment, is a 20-item, 4-point Likert-type scale (1 Not at all, 2 A little, 3 A lot, 4 Completely) that indicates the frequency of the feelings and behaviors expressed by the individual. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 in the state anxiety scale contain reversed statements. The scale is scored by adding 50 points to the difference between the total weighted scores of the direct statements and the reverse statements. Accordingly, the lowest score that can be obtained from the scale is 20, and the highest score is 80. An increase in the score obtained from the scale indicates that state anxiety has developed. A score below 36 on the scale indicates no anxiety, a score between 37-42 indicates mild anxiety, and a score of 42 and above indicates high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Ammochostos, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie W, Ye F, Yan X, Cao M, Ho MH, Kwok JYY, Lee JJ. Acupressure can reduce preoperative anxiety in adults with elective surgery: A systematic review and meta-analysis of randomised controlled trials. Int J Nurs Stud. 2023 Sep;145:104531. doi: 10.1016/j.ijnurstu.2023.104531. Epub 2023 May 22. PMID 37321140
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37321140/